CLINICAL TRIAL: NCT07119684
Title: The Effect of Duration and Frequency of Walking Exercise on Cognitive Functions: A Randomized Controlled Comparative Study
Brief Title: The Effect of Duration and Frequency of Walking Exercise on Cognitive Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Zeynep Tuna, associate professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: cognitiveshamelGazi
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Cognitive Function and Well-Being; Healthy Participants; Walking
Keywords: Exercise Duration, Exercise Frequency, Cognitive Function, Walking Exercise

STUDY DESIGN:
Intervention Model Description: Two groups (10-minute walking group vs. 30-minute walking group)
  Each group receives a different intervention
  Participants stay in the same group throughout the study (no crossover)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants were not blinded (they knew their group)
  Investigators (those conducting and monitoring the intervention) were blinded
  Outcomes assessors (evaluating cognitive tests) were blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short-Duration Walking Group (Experimental): Participants walked 3 sessions of 10 minutes per day, five days a week for 6 weeks, at 60% of their maximum heart rate.
  Interventions: Behavioral: Short-Duration Walking Exercise
- Long-Duration Walking Group (Active Comparator): Participants walked 1 continuous 30-minute session per day, five days a week for 6 weeks, at 60% of their maximum heart rate.
  Interventions: Behavioral: Long-Duration Walking Exercise

INTERVENTIONS:
Behavioral: Short-Duration Walking Exercise — articipants performed three 10-minute walking sessions per day, 5 days per week for 6 weeks, at 60% of their maximum heart rate on a treadmill.
  Arms: Short-Duration Walking Group
Behavioral: Long-Duration Walking Exercise — Participants performed one continuous 30-minute walking session per day, 5 days per week for 6 weeks, at 60% of their maximum heart rate on a treadmill.
  Arms: Long-Duration Walking Group

SUMMARY:
Physical activity is very important for staying healthy and improving how well our brain works. Walking is a simple and easy way to exercise that can help people of all ages feel better physically and mentally. It's affordable, easy to do, and doesn't require special equipment. Walking can improve memory, thinking speed, and problem-solving skills, which are important for everyday life.

This study looks at whether doing shorter walks more often (like three 10-minute walks a day) is as good for the brain as doing one longer walk (one 30-minute walk a day). This is important because many people find it hard to fit long exercise sessions into their day due to busy schedules, health issues, or personal preferences.

By understanding which way of walking helps the brain the most, doctors and patients can choose exercise plans that are easier to stick to and still improve thinking skills. This study will compare these two walking routines over 6 weeks to see how they affect brain health.

This clinical trial investigates the cognitive effects of two different walking exercise protocols over a 6-week period. Participants will either complete three daily 10-minute walking sessions or a single continuous 30-minute walking session. The study aims to determine whether shorter, more frequent exercise sessions provide cognitive benefits comparable to a longer, single session. Outcomes will focus on improvements in memory, processing speed, and executive function. Findings will inform recommendations for accessible and flexible exercise programs to enhance cognitive health.

ELIGIBILITY:
Inclusion Criteria:

* Female

Aged between 18 and 25 years

Sedentary lifestyle, defined as taking <5000 steps/day in the previous week

Non-smoker

Having a work or school schedule that allows consistent participation in the 6-week walking program

Able to walk on a treadmill

Provided written informed consent

Exclusion Criteria:

* Body Mass Index (BMI) ≥ 30 kg/m²

Participation in another regular exercise program during the study period

Neurological conditions (e.g., stroke, epilepsy)

Severe cardiovascular conditions (e.g., heart failure, arrhythmias)

Any physical limitation that prevents safe walking on a treadmill

Pregnancy

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
Change in Digit Symbol Substitution Test (DSST) Score | Baseline and 6 weeks post-intervention
  Main endpoint; large effect size; reflects executive function & speed

SECONDARY OUTCOMES:
Change in Stroop Test | Baseline and 6 weeks post-intervention
  Exploring other areas the intervention might influence (e.g., different aspects of cognitive function).

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Demographic data: age, height, weight, BMI
  Group assignment: 10-minute or 30-minute walking group
  Cognitive test scores:
  Stroop Test Word (STW)
  Stroop Test Color (STC)
  Stroop Test Word-Color (STWC)
  Digit Symbol Substitution Test (DSST)
  Pre- and post-intervention scores for all cognitive assessments
Supporting Information: SAP

DOCUMENTS (1):
  • Study Protocol (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/84/NCT07119684/Prot_000.pdf